CLINICAL TRIAL: NCT06332326
Title: Investigation of the Efficacy of Non-Invasive Vagus Nerve Stimulation and Physiotherapy in Unilateral Vestibular Hypofunction Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Tugba Turk Kalkan, principal investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E-10840098-772.02-4966
Record Dates: First submitted 2024-03-14; First posted 2024-03-27 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Vestibular Diseases; Vestibular Vertigo; Vertigo
Keywords: unilateral vestibular hypofunction; Non-Invasive Vagus Nerve Stimulation; balance; vestibular rehabilitation
MeSH Terms: conditions — Vestibular Diseases; Vertigo

STUDY DESIGN:
Intervention Model Description: 40 patients diagnosed with UHV were included. Patients were randomized into 2 separate groups (20 people in the vestibular rehabilitation group, 20 people in the vagus nerve stimulation group in addition to vestibular rehabilitation).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR+VAGUS GROUP (Experimental): VR+VAGUS GROUP (n=20): PATIENTS USED NON-INVASIVE VAGUS NERVE STIMULATION IN ADDITION TO VESTIBULAR REHABILITATION
  Interventions: Device: non-invasive vagus nerve stimulation; Behavioral: vestibular rehabilitation
- VR GROUP (Active Comparator): VR GROUP (n=20) : PATİENTS UNDERGOİNG VESTİBULAR REHABİLİTATİON
  Interventions: Behavioral: vestibular rehabilitation

INTERVENTIONS:
Device: non-invasive vagus nerve stimulation — non-invasive vagus nerve stimulation: patients will receive non-invasive vagus nerve stimulation.
  Arms: VR+VAGUS GROUP
Behavioral: vestibular rehabilitation — vestibular rehabilitation: Patients will be given specially structured vestibular rehabilitation exercises.

SUMMARY:
The purpose of this study: To investigate the effectiveness of non-invasive vagus nerve stimulation and vestibular rehabilitation applications in patients diagnosed with Unilateral Vestibular Hypofunction (UVH).

DETAILED DESCRIPTION:
It was planned to include 40 patients diagnosed with UHV in the study. Patients were randomized into 2 separate groups (20 people in the vestibular rehabilitation group, 20 people in the vagus nerve stimulation group in addition to vestibular rehabilitation).

ELIGIBILITY:
Inclusion Criteria:

* He learned about unilateral peripheral vestibular hypofunction with videonystagmography
* Being able to communicate well

Exclusion Criteria:

* Having cognitive impairment
* Presence of central neurological disease
* Lack of cooperation
* Previous ear surgery
* Accompanied by Benign Proxysmal Positional Vertigo
* Having acute Meniere's disease
* Finding pathology in temporal bone MRI
* Having a lower extremity disorder that prevents walking
* Evidence of central pathology in videonystagmography results

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Modified-CTSIB | 30 minutes
  Modified-CTSIB; It is generally used as a semi-quantitative test measurement and clinical practice in which points are scored based on the ability to perform various standing static positions It is a test. It covers different situations where the patient must stand under different conditions: foam surface versus hard floor, tested with eyes open and closed in six different test groups.
Semitandem test | 10 minutes
  semitandem stance positions; The conditions (sec) of remaining in balance with eyes open and closed on hard and soft surfaces will be measured.
tandem test | 10 minutes
  tandem semitandem stance positions; The conditions (sec) of remaining in balance with eyes open and closed on hard and soft surfaces will be measured.
one-leg standing test | 10 minutes
  one-leg standing test; The conditions (sec) of remaining in balance with eyes open and closed on hard and soft surfaces will be measured.
Unterberger test | 5 minutes
  Unterberger test: The patient first takes 10 steps quickly with his eyes open, then With his eyes closed, he takes 50 steps quickly in place. If there is a lesion, apply it to the side of the lesion.
  correct deviation occurs.
VAS Visual Analogue Scale (dizziness severity) | 5 minutes
  Visual Analogue Scale will be applied to evaluate dizziness severity and patient satisfaction. With this scale, scoring from 0 to 10 is requested. While 0 indicates the lowest dizziness severity and lowest patient satisfaction, 10 indicates the highest dizziness severity and highest patient satisfaction.
Dynamic visual acuity test | 5 minutes
  Dynamic visual acuity test; It measures the ability to see an object during rapid head movements.

SECONDARY OUTCOMES:
Dizziness Handicap Inventory Scale | 5 minutes
  It was developed to measure disability in patients complaining of dizziness and imbalance and is used in treatment follow-up. It is a survey consisting of 25 questions about the patient's physical (7 questions), functional (9 questions) and emotional (9 questions) status, and which patients can apply themselves in line with their complaints. Patients rate the questions as 0 (no), 2 (sometimes) and 4 (yes) based on their complaints. high scores describe severe dizziness.
Tampa Kinesiophobia Scale | 5 minutes
  The Tampa Kinesiophobia Scale will be used to evaluate kinesiophobia. It is a 17-question scale developed to measure fear of injury. The scale includes injury/re-injury and fear-avoidance parameters in work-related activities. High scores describe severe kinesiophobia.
Hospital Anxiety and Depression Scale (HAD) | 5 minutes
  The Tampa Kinesiophobia Scale will be used to evaluate kinesiophobia. It is a 17-question scale developed to measure fear of injury. The scale includes injury/re-injury and fear-avoidance parameters in work-related activities. High scores describe higher levels of depression and anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: tuğba türk kalkan, MD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)